CLINICAL TRIAL: NCT02409550
Title: CARATKids: Italian Validation of Asthma and Allergic Rhinitis Control Test in Children
Status: Completed | Type: Observational
Sponsor: Stefania La Grutta, MD (Other)
Responsible Party: Sponsor-Investigator, Stefania La Grutta, MD, Stefania La Grutta, MD. Senior Researcher. Coordinator of Pediatric Allergy and Asthma Research Group. Institute of Biomedicine and Molecular Immunology, IBIM, National Research Council of Palermo, Italy., Istituto per la Ricerca e l'Innovazione Biomedica
Organization: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Other Study IDs: 11/2014
Record Dates: First submitted 2015-03-24; First posted 2015-04-07 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Allergic Rhinitis; Asthma
Keywords: Allergic Rhinitis; Asthma; Children; Control
MeSH Terms: conditions — Rhinitis, Allergic; Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 113 patients with concomitant asthma and allergic rhinitis: 113 patients with concomitant asthma and allergic rhinitis followed up from at least 3 months will be enrolled for the validation process at outpatient clinic of Pediatric Allergology & Pulmonology (PAP) of Respiratory Disease Research Center (RDRC) within the Institute of Biomedicine and Molecular Immunology (IBIM) of the National Research Council (CNR) of Palermo (RDRC-IBIM CNR), Italy.
  Interventions: Other: CARATKids Questionnaire

INTERVENTIONS:
Other: CARATKids Questionnaire

SUMMARY:
This project is an observational study for the Italian language validation of the CARATKids questionnaire investigating the asthma and coexisting allergic rhinitis control in children. 113 patients with concomitant asthma and allergic rhinitis followed up from at least 3 months will be enrolled for the validation process at outpatient clinic of Pediatric Allergology & Pulmonology (PAP) of Respiratory Disease Research Center (RDRC) within the Institute of Biomedicine and Molecular Immunology (IBIM) of the National Research Council (CNR) of Palermo (RDRC-IBIM CNR), Italy.

The study will be completed in two medical examination, within 3-6 weeks of each other.

CARATKids questionnaire, VAS (Visual Analogic Scale) and C-ACT (Children Asthma Control Test) will be filled by each patient.

The main outcome is the Italian language validation of the CARATKids questionnaire investigating the coexisting asthma and allergic rhinitis control in children.

ELIGIBILITY:
Inclusion Criteria:

* 113 patients with concomitant asthma and allergic rhinitis followed up from at least 3 months
* 12 < years old > 6

Exclusion Criteria:

* Patients with asthma only or allergic rhinitis only, or younger or older than the targeted age group

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 113 patients with concomitant asthma and allergic rhinitis followed up from at least 3 months will be enrolled for the validation process at outpatient clinic of Pediatric Allergology & Pulmonology (PAP) of Respiratory Disease Research Center (RDRC) within the Institute of Biomedicine and Molecular Immunology (IBIM) of the National Research Council (CNR) of Palermo (RDRC-IBIM CNR), Italy.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
CARATKids Italian language validation | 3 weeks
  The main objective of the study is the assessment process of the tool CARATKids, in a scholastic children Italian population affected by coexisting asthma and allergic rhinitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Biomedicine and Molecular Immunology, IBIM, Palermo, Palermo, Italy

IPD SHARING:
Plan to Share IPD: Yes
The IPD collected will be available on May 2016.
  The following participant data will be shared:
  * Asthma severity level
  * Asthma control level
  * Pulmonary function tests
  * Demographic characteristics All IPD will be obtained from statistical analysis on the dedicated database in which all data are stored.